CLINICAL TRIAL: NCT06863168
Title: Effective Cigarillo Public Education Messaging for Black Young Adults
Brief Title: Cigarillo Public Education Messaging for Black Young Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2307010033; R00CA272919 (NIH)
Record Dates: First submitted 2025-03-03; First posted 2025-03-07 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cigarillo Smoking

STUDY DESIGN:
Intervention Model Description: The intervention consists of cigarillo public education messages that will be delivered online for four days each week for four weeks. Messages will communicate the health harm and nicotine addiction risks of cigarillo smoking alone (i.e., long-term health risks, short-term health risks, social health risks, nicotine addiction); or, contextualized to outcome expectancies of cigarillo smoking sensory experience, anticipated pleasure, relaxation, and satisfaction from cigarillo smoking, social persona/admiration related to cigarillo smoking, and that smoking does not align with personal values and authenticity. These intervention messages will be compared to a control messaging arm. Messaging order of the 16 messages per study arm will be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Non-Tobacco Messages (No Intervention): Participants in the control arm will receive messages about food safety. Four of the 16 total messages will be emailed with a survey link on four days each week for four weeks.
- Cigarillo Harm Messaging (Experimental): Participants in the harm messaging arm will receive messages about the 1) long-term health risks, 2) short-term health risks, 3) social health risks, and 4) nicotine addiction of cigarillo smoking. Four of the 16 total messages will be emailed with a survey link on four days each week for four weeks. Each week's 4 messages will be randomized and include one message from the four harm themes.
  Interventions: Behavioral: Cigarillo Health Harm and Nicotine Addiction Messaging
- Cigarillo Harm Messages Contextualized to Outcome Expectancies (Experimental): Participants in the harm messaging contextualized to outcome expectancies arm will receive messages about the health harm and nicotine addiction risks of cigarillo smoking contextualized to one of the following themes: 1) smoking sensory experience, 2) anticipated pleasure, relaxation, and satisfaction from smoking, 3) social persona/admiration related to smoking, and 4) that smoking does not align with personal values and authenticity. Four of the 16 total messages will be emailed with a survey link on four days each week for four weeks. Each week's 4 messages will be randomized and include one message from the four harm themes.
  Interventions: Behavioral: Cigarillo Health Harm and Nicotine Addiction Messaging Contextualized to Outcome Expectancies

INTERVENTIONS:
Behavioral: Cigarillo Health Harm and Nicotine Addiction Messaging — Participants in the harm messaging arm will receive messages about the 1) long-term health risks, 2) short-term health risks, 3) social health risks, and 4) nicotine addiction of cigarillo smoking.
  Arms: Cigarillo Harm Messaging
Behavioral: Cigarillo Health Harm and Nicotine Addiction Messaging Contextualized to Outcome Expectancies — Participants in the harm messaging contextualized to outcome expectancies arm will receive messages about the health harm and nicotine addiction risks of cigarillo smoking (i.e., 1) long-term health risks, 2) short-term health risks, 3) social health risks, and 4) nicotine addiction of cigarillo smoking) contextualized to one of the following themes: 1) smoking sensory experience, 2) anticipated pleasure, relaxation, and satisfaction from smoking, 3) social persona/admiration related to smoking, and 4) that smoking does not align with personal values and authenticity.
  Arms: Cigarillo Harm Messages Contextualized to Outcome Expectancies

SUMMARY:
This is a 3-arm randomized controlled trial to examine the effects of cigarillo public education messages among Black young adults who are at-risk for established cigarillo smoking. The primary outcomes are cigarillo harm perceptions, outcome expectancies, and use intentions at 3-month follow-up. Exploratory outcomes are use behaviors (cigarillo smoking initiation and use behaviors) measured at 3-month follow-up. These outcomes will also be measured at 1-month follow-up time point.

DETAILED DESCRIPTION:
This is a 3-arm randomized controlled trial to examine the effects of cigarillo public education messages among Black young adults who are at-risk for established cigarillo smoking. The primary outcomes are cigarillo harm perceptions, outcome expectancies, and use intentions at 3-month follow-up. Exploratory outcomes are use behaviors (cigarillo smoking initiation and use behaviors) measured at 3-month follow-up. These outcomes will also be measured at 1-month follow-up time point. Participants will be recruited online through research panel services. Eligible participants will be those who: 1) are of non-Hispanic Black or African American ethnicity and race, respectively; 2) are between 18 to 30 years of age; 3) have never used cigarillos fairly regularly but are deemed susceptible to cigarillo smoking or currently smokes cigarillos some days but not every day; and 4) have no history of fairly regular use of any other tobacco products (i.e., little cigars, large cigars, cigarettes, hookah tobacco, electronic vaping products, smokeless tobacco, and heated tobacco products). Potential participants will be provided with a brief description of the study and a link to the eligibility screener. Those who are eligible will proceed to the online consent form. Eligible and consenting participants will complete an online assessment of demographic characteristics, tobacco use intentions and behaviors, attitudes, and perceptions (e.g., harm perceptions, outcome expectancies), alcohol use, cannabis use, and life experiences. After completing the baseline assessment, participants will be randomly assigned in approximately equal numbers into one of three study arms: 1) cigarillo harm messaging alone; 2) cigarillo harm messaging contextualized to outcome expectancies; and 3) control messaging arm. Each arm includes 16 messages. Harm messaging includes messages about the risks of cigarillo smoking including long-term health risks, short-term health risks, social health risks, and nicotine addiction. Harm messaging contextualized with outcome expectancies includes messages about the health harm and nicotine addiction risks of cigarillos contextualized to cigarillo smoking sensory experiences, anticipated pleasure, relaxation, and satisfaction from cigarillo smoking, social persona/admiration related to cigarillo smoking, and that cigarillo smoking does not align with personal values and authenticity. Control messaging includes messages about food safety. Participants will be emailed and asked to view four study arm messages (i.e., one message per theme) on four days each week for four weeks. On the 4th day of each week, participants will also complete measures of message responses for the four messages viewed that day. Following the intervention period, message recall, tobacco use intentions and behaviors, attitudes, perceptions (e.g., harm perceptions, outcome expectancies), alcohol use, and cannabis use will be assessed at 1-month and 3-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Be between 18 to 30 years of age;
* Self-identify as non-Hispanic Black or African American ethnicity and race, respectively;
* Must be able to communicate, read, and write in the English language;
* Have never used cigarillos fairly regularly based on a valid measure but are deemed susceptible to cigarillo smoking based on a valid 4-item susceptibility measure; OR currently smokes cigarillos some days but not every day (i.e., experimentation)
* And must have no history of fairly regular use of any other tobacco products (i.e., little cigars, large cigars, cigarettes, hookah tobacco, electronic vaping products, smokeless tobacco, and heated tobacco products)

Exclusion Criteria:

* Persons who are younger than 18 years of age or older than 30 years of age.
* Persons who do not self-identify as a non-Hispanic Black/African American person.
* Persons who are not deemed susceptible based on a valid susceptibility measure (i.e., not susceptible to cigarillo smoking)
* Persons who have fairly regular use of any tobacco product (i.e., persons with a former or current established pattern of any tobacco use including cigarillos, little cigars, large cigars, cigarettes, hookah tobacco, electronic vaping products, smokeless tobacco, and heated tobacco products)
* Persons who are unable to read, write, and communicate in English language. The informed consent and other materials, including surveys, are only available in the English language for this study. Additionally, trained staff members that will communicate and interact with participants for this study can only speak in English.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Estimated)
Dates: Start 2025-04-17 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Cigarillo harm perceptions | 1-month; 3-month
  Cigarillo absolute harm perceptions will be measured using three self-report items. One item assesses perceptions of how harmful cigarillo smoking is (1=not at all harmful to 5=extremely harmful). Another item assesses perceptions of likelihood of addiction (1=not likely to 5=very likely). A multi-item measure will measure the level of agreement (1=strongly disagree to 5=strongly agree) that cigarillo smoking would cause various health harms and nicotine addiction risks.
Cigarillo outcome expectancies | 1-month; 3-month
  Cigarillo outcome expectancies will be measured via level of agreement (1=strongly disagree to 5=strongly agree) with various statements of potential anticipated outcomes from cigarillo smoking.
Cigarillo use intentions | 1-month; 3-month
  Cigarillo use intentions will be measured using self-report items related to cigarillo smoking susceptibility (i.e., Do you think that you will use a cigarillo soon?; Do you think that you will use a cigarillo in the next year?; Do you think that in the future you might experiment with cigarillos?; If one of your best friends were to offer you a cigarillo, would you smoke it?) with response options including "definitely yes"; "probably yes"; "probably not"; and "definitely not". Combination of responses other than "definitely not" to all four items will be considered susceptible to cigarillo smoking. Cigarillo use intentions will also be assessed by one's willingness to smoke cigarillos in various situations with responses ranging from unwilling=0% to extremely willing=100%.

SECONDARY OUTCOMES:
Cigarillo use behaviors | 1-month; 3-month
  Cigarillo use behaviors will be measured by assessing cigarillo smoking initiation (Have you smoked a cigarillo, even one or two puffs?) and use behaviors (e.g., fairly regular use, current use some days or everyday, the last time a cigarillo was smoked, and the number of cigarillos smoked in the past 30 days) from the baseline time-point.

CONTACTS AND LOCATIONS:
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No